CLINICAL TRIAL: NCT02612779
Title: A Phase 2, Multiple Cohort Study of Elotuzumab in Combination With Pomalidomide and Low-Dose Dexamethasone (EPd), and in Combination With Nivolumab (EN), in Patients With Multiple Myeloma Relapsed or Refractory to Prior Treatment With Lenalidomide.
Brief Title: A Study of Elotuzumab in Combination With Pomalidomide and Low Dose Dexamethasone and Elotuzumab in Combination With Nivolumab in Patients With Multiple Myeloma Relapsed or Refractory to Prior Treatment With Lenalidomide.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA204-142
Record Dates: First submitted 2015-11-20; First posted 2015-11-24 (Estimated); Results first posted 2020-08-06 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — elotuzumab; pomalidomide; Dexamethasone; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Elotuzumab + Pomalidamide + Low Dose Dexamethasone (EPd) (Experimental): patients will receive treatment with elotuzumab in combination with pomalidomide and low-dose dexamethasone. Patients are eligible to receive Nivolumab at progression.
  Interventions: Drug: Elotuzumab; Drug: Pomalidomide; Drug: Dexamethasone; Drug: Nivolumab
- Elotuzumab + Nivolumab (EN) (Experimental): Patients will receive treatment with a combination of elotuzumab and nivolumab
  Interventions: Drug: Elotuzumab; Drug: Nivolumab

INTERVENTIONS:
Drug: Elotuzumab
Drug: Pomalidomide
  Arms: Elotuzumab + Pomalidamide + Low Dose Dexamethasone (EPd)
Drug: Dexamethasone
  Arms: Elotuzumab + Pomalidamide + Low Dose Dexamethasone (EPd)
Drug: Nivolumab

SUMMARY:
Study of elotuzumab in combination with pomalidomide and low dose dexamethasone (EPd Cohort) and elotuzumab in combination with nivolumab (EN Cohort) to assess the safety and efficacy of these combination therapies for treatment of relapsed or refractory MM patients.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

1. All subjects must have documented disease progression per IMWG criteria during or after their last anti-myeloma therapy.
2. ECOG Performance Status less than or equal to 2
3. Subject Re-enrollment: This study permits the re-enrollment of a subject that has discontinued the study as a pre-treatment failure (ie, has not been treated). If re-enrolled, the subject must be re-consented.
4. EPd Cohort:

   * must have received at least 1 but no greater than 2 prior lines of therapy (note: induction and stem cell transplants with or without maintenance therapy is considered 1 line of therapy)
   * Subjects must have received prior treatment with a lenalidomide-containing regimen for at least 2 consecutive cycles (full therapeutic dose) and must have been deemed as relapsed, refractory, or intolerant. Refractory is defined as progressing on-treatment or within 60 days of the last dose.
5. EN Cohort:

   * Subjects must have received at least 3 prior lines of therapy including a proteasome inhibitor (PI) and an immunomodulatory (IMID) agent OR were double-refractory to both an IMID and a PI. Refractory is defined as progressing on-treatment or within 60 days of the last dose.

Exclusion Criteria:

1. Subjects with solitary bone or extramedullary plasmacytoma as the only evidence of plasma cells dyscrasia
2. Subjects with monoclonal gammopathy of undetermined significance (MGUS), smoldering multiple myeloma (SMM), primary amyloidosis, Waldenstrom's macroglobulinemia, or POEMS syndrome (plasma cell dyscrasia with poly neuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
3. Subjects with Central Nervous System involvement with multiple myeloma

Other protocol defined inclusion/exclusion criteria could apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2016-02-09 (Actual); Primary Completion 2019-07-29 (Actual); Study Completion 2020-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (22):
- United States (22):
  - Southern Cancer Center, Mobile, Alabama
  - Sansum Clinic - USOR, Santa Barbara, California
  - Colorado Blood Cancer Institute - PPDS, Denver, Colorado
  - Rocky Mountain Cancer Centers (Williams) - USOR, Denver, Colorado
  - Florida Cancer Specialists - EAST - SCRI - PPDS, St. Petersburg, Florida
  - Florida Cancer Specialists - NORTH - SCRI - PPDS, St. Petersburg, Florida
  - Illinois Cancer Care, Peoria, Illinois
  - American Oncology Partners of Maryland, PA, Bethesda, Maryland
  - Bay Hematology Oncology, Easton, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Center, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - Mount Sinai Medical Center, New York, New York
  - Greenville Health System, Greenville, South Carolina
  - Avera Health Care, Sioux Falls, South Dakota
  - Jones Clinic PC, Germantown, Tennessee
  - Tennessee Oncology NASH - SCRI - PPDS, Nashville, Tennessee
  - Texas Oncology (Loop) - USOR, San Antonio, Texas
  - Virginia Cancer Specialists (Leesburg) - USOR, Leesburg, Virginia
  - Swedish Medical Center, Seattle, Washington
  - Cancer Care Northwest, Spokane Valley, Washington
  - Aurora Health Care, Burlington, Wisconsin

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: EPd cohort: 68 participants entered the treatment period. EN cohort: 6 participants entered the treatment period.
Groups:
- EPd Cohort: Participants received treatment with Elotuzumab in combination with Pomalidomide and low-dose Dexamethasone in a 28 day cycle.
- EN Cohort: Participants received Elotuzumab in combination with Nivolumab in a 28-day cycle.
Period: Overall Study
Arm/Group | EPd Cohort | EN Cohort
Started | 68 | 6
Completed | 0 | 0
Not Completed | 68 | 6
Not completed — Administrative reason by sponsor | 4 | 1
Not completed — No longer meet study criteria | 0 | 1
Not completed — Disease progression | 29 | 2
Not completed — Study drug toxicity | 10 | 1
Not completed — Death | 1 | 0
Not completed — Adverse event unrelated to study drug | 5 | 0
Not completed — Participant withdrew consent | 4 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Maximum clinical benefit | 10 | 1
Not completed — Other reasons | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EPd Cohort | EN Cohort | Total
Number analyzed (Participants) | 68 | 6 | 74
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.3 (9.11) | 69.5 (10.56) | 65.6 (9.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 3 | 36
  Male | 35 | 3 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 0 | 6
  Not Hispanic or Latino | 61 | 6 | 67
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian1 | 1 | 0 | 1
  Black or African American | 4 | 3 | 7
  White | 58 | 3 | 61
  Other | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from first dosing date to the date of the first documented progression or death due to any cause, whichever occurs first.
  Progression is determined per International Myeloma Working Group (IMWG) uniform criteria.
  Participants who die without a reported prior progression were considered to have progressed on the date of their death.
  Participants who did not progress or die were censored on the date of their last evaluable assessment. Participants who did not have any on study efficacy assessments and did not die were censored on the first dosing date.
  Participants who switched to subsequent therapy prior to documented progression were censored on the date of the last evaluable assessment prior to the initiation of the new therapy.
Time Frame: From first dose to study completion date (up to approximately 50 months)
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | EPd Cohort
Number analyzed (Participants) | 68
Months | 11.1 [7.4 to 15.0]

2. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percent of participants with best overall response of partial response (PR) or better. Response is determined per IMWG uniform criteria.
Time Frame: From first dose to study completion date (up to approximately 50 months)
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | EN Cohort
Number analyzed (Participants) | 6
Percent of Participants | 16.7 [0.42 to 64.12]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: as for outcome 2
Time Frame: From first dose to study completion date (up to approximately 50 months)
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | EPd Cohort
Number analyzed (Participants) | 68
Percent of Participants | 51.5 [39.03 to 63.78]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: as for outcome 1
Time Frame: From first dose to study completion date (up to approximately 50 months)
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | EN Cohort
Number analyzed (Participants) | 6
Months | 1.9 [0.6 to NA] — Upper limit not estimable

5. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from first dosing date to the date of death from any cause.
Time Frame: From first dose to study completion date (up to approximately 50 months)
Population: All treated participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | EPd Cohort | EN Cohort
Number analyzed (Participants) | 68 | 6
Months | 41.2 [22.7 to NA] — Upper limit not estimable | NA [0.6 to NA] — The median was not reached because of an insufficient number of events

ADVERSE EVENTS:
Time Frame: From first dose to 100 days after last dose
Arm/Group | EPd Cohort | EN Cohort
All-Cause Mortality (participants affected / at risk) | 32/68 | 2/6
Serious Adverse Events (participants affected / at risk) | 39/68 | 3/6
Other Adverse Events (participants affected / at risk) | 66/68 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EPd Cohort (N=68) | EN Cohort (N=6)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0
Cardiac arrest (Cardiac disorders) | 2 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Amaurosis fugax (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Disease progression (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Appendicitis perforated (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 4 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Herpes simplex encephalitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Klebsiella bacteraemia (Infections and infestations) | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 18 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0
Salmonella bacteraemia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 3 | 0
Septic shock (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 4 | 0
Urosepsis (Infections and infestations) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Vascular access site bruising (Injury, poisoning and procedural complications) | 1 | 0
Influenza B virus test positive (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EPd Cohort (N=68) | EN Cohort (N=6)
Anaemia (Blood and lymphatic system disorders) | 15 | 2
Leukopenia (Blood and lymphatic system disorders) | 13 | 0
Lymphopenia (Blood and lymphatic system disorders) | 11 | 1
Neutropenia (Blood and lymphatic system disorders) | 24 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 1
Cataract (Eye disorders) | 5 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 5 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 17 | 1
Diarrhoea (Gastrointestinal disorders) | 24 | 0
Dyspepsia (Gastrointestinal disorders) | 4 | 1
Nausea (Gastrointestinal disorders) | 14 | 2
Stomatitis (Gastrointestinal disorders) | 3 | 1
Toothache (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 7 | 0
Chills (General disorders) | 4 | 0
Fatigue (General disorders) | 37 | 1
Feeling jittery (General disorders) | 4 | 0
Oedema peripheral (General disorders) | 17 | 0
Pyrexia (General disorders) | 10 | 1
Bronchitis (Infections and infestations) | 4 | 0
Cellulitis (Infections and infestations) | 6 | 0
Conjunctivitis (Infections and infestations) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 6 | 0
Pneumonia (Infections and infestations) | 4 | 0
Sinusitis (Infections and infestations) | 5 | 0
Upper respiratory tract infection (Infections and infestations) | 25 | 0
Contusion (Injury, poisoning and procedural complications) | 4 | 0
Fall (Injury, poisoning and procedural complications) | 7 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 4 | 2
Neutrophil count decreased (Investigations) | 7 | 0
Weight decreased (Investigations) | 5 | 0
Weight increased (Investigations) | 7 | 0
Decreased appetite (Metabolism and nutrition disorders) | 13 | 2
Dehydration (Metabolism and nutrition disorders) | 7 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 4 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 10 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 17 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 0
Dizziness (Nervous system disorders) | 9 | 1
Dysgeusia (Nervous system disorders) | 4 | 0
Headache (Nervous system disorders) | 11 | 1
Hypoaesthesia (Nervous system disorders) | 4 | 0
Neuropathy peripheral (Nervous system disorders) | 4 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 6 | 0
Syncope (Nervous system disorders) | 4 | 0
Tremor (Nervous system disorders) | 6 | 0
Anxiety (Psychiatric disorders) | 7 | 0
Depression (Psychiatric disorders) | 7 | 0
Insomnia (Psychiatric disorders) | 14 | 1
Dysuria (Renal and urinary disorders) | 5 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 22 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 6 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 2 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 4 | 0
Flushing (Vascular disorders) | 4 | 1
Hot flush (Vascular disorders) | 4 | 0
Hypertension (Vascular disorders) | 8 | 0
Hypotension (Vascular disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2018-03-08): https://cdn.clinicaltrials.gov/large-docs/79/NCT02612779/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-24): https://cdn.clinicaltrials.gov/large-docs/79/NCT02612779/SAP_001.pdf